CLINICAL TRIAL: NCT00222508
Title: Microvascular Complications of Cystic Fibrosis Related Diabetes
Brief Title: The Microvascular Complications Study
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: Cystic Fibrosis Foundation (Other); Vikings Children Fund (Unknown); Moran, Antoinette, M.D. (Individual)
Responsible Party: Sponsor
Other Study IDs: 0012M75862
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-07

CONDITIONS: Cystic Fibrosis Related Diabetes
Keywords: Cystic Fibrosis; Diabetes; Complications
MeSH Terms: conditions — Cystic Fibrosis; Diabetes Mellitus

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Our general aim is to determine the prevalence of diabetic microvascular complications in CFRD patients with and without fasting hyperglycemia, and to explore whether the presence of these complications is related to diabetes or CF factors. This cross-sectional study will provide pilot data for a longitudinal study of diabetes complications in CF.

DETAILED DESCRIPTION:
Microvascular complications of diabetes such as eye, kidney and nerve disease are common in individuals with type 1 and type 2 diabetes, and are a source of significant morbidity and mortality. Microvascular diabetes complications have been anecdotally reported in cystic fibrosis related diabetes (CFRD), but their prevalence is unknown. 40% of adult CF patients have CFRD, which shares features of both type 1 and type 2 diabetes but is a distinct clinical entity (1). Many clinicians are reluctant to add the burden of aggressive diabetes management to the already complex medical regimen of these patients. It is sometimes stated that they will not live long enough to develop complications of diabetes. However, longevity in CF has dramatically increased, and many patients now live into their thirties, forties, and fifties. As they live longer, it becomes increasingly likely that at least some will develop diabetes complications. A better understanding of this negative outcome would help resolve the question of whether aggressive screening and management of diabetes is necessary in CF.

As in other forms of diabetes, duration of diabetes and the magnitude of chronic hyperglycemia are probably important determinants of microvascular complications in CFRD. This information is not usually known at the time of presentation of CFRD because of the insidious onset of the disease. Theoretically, CF pulmonary disease, including chronic hypoxia and venous congestion related to pulmonary hypertension, may additionally aggravate microvascular changes. However, the metabolic differences between CFRD and type 1 and type 2 diabetes may also serve to protect CF patients from some diabetes complications. At the time diabetes complications develop, patients with type 1 and type 2 diabetes tend to have concomitant obesity, hypertension, insulin resistance, hyperlipidemia and atherosclerotic cardiovascular disease. These factors, which are generally absent in CF, may contribute to the pathophysiology of microvascular complications in other forms of diabetes.

The University of Minnesota CF Center is in the unique position of having a well-characterized diabetes population, since diabetes screening was instituted several years ago as part of routine annual CF studies. In our population of 450 CF patients, 113 have been diagnosed with diabetes, and the remainder are known to have either normal or impaired glucose tolerance. In addition to our CFRD experience, the University of Minnesota has a strong background of experience in large population-based screening and intervention trials concerning diabetes complications. Not only were we a participating center in the NIH-sponsored multi-center Diabetes Control and Complications Trial (DCCT) (2) and the current DCCT follow-up Epidemiology of Diabetes Interventions and Complications trial (EDIC), but our laboratory was central reference laboratory for the DCCT and EDIC. Thus, our physicians, nurses, biostatisticians, GCRC staff and laboratory staff are all quite knowledgeable and experienced in the methods to be used in the present application.

ELIGIBILITY:
Inclusion Criteria:

CFRD patients with and without fasting hyperglycemia

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: CFRD Patients
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2001-04; Study Completion 2005-07

CONTACTS AND LOCATIONS:
Overall Officials: Antoinette Moran, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States